CLINICAL TRIAL: NCT06813209
Title: Effects of Transcranial Electrical Stimulation by Continuous Current on the Right and Left Dorsolateral Prefrontal Cortex Associated or Not with Non-invasive Vagus Nerve Stimulation in Adult Individuals with Chronic Stress
Brief Title: Effects of Transcranial Electrical Stimulation in Chronic Stress
Acronym: NEUROSTIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Collaborators: Universidade Federal de Alfenas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1328
Record Dates: First submitted 2024-12-05; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-12

CONDITIONS: Stress; Sleep
Keywords: Transcranial electrical stimulation by direct current; tDCS; non-invasive vagus nerve stimulation; stress; tVNS
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- tDCS True Modulation (Experimental): Participants will be delivered true treatment for 20 minutes each session
  Interventions: Device: tDCS
- tDCS Sham group (Sham Comparator): Sham group will be delivers a simulated treatment; the current will be applied for only 60 seconds, with the setup remaining in place for 20 minutes.
  Interventions: Device: tDCS
- tVNS True (Experimental): For true tVNS stimulation, the technique will be performed with the electrodes positioned on the upper concha of the left ear, using gel for better current distribution.
  Interventions: Device: tVNS
- tVNS Sham (Sham Comparator): For sham tVNS stimulation, the technique will be performed in the same way as true stimulation; however, the device will be programmed to deliver 0 Hz.
  Interventions: Device: tVNS

INTERVENTIONS:
Device: tDCS — For true tDCS, the technique will be performed with the anode over the right dorsolateral prefrontal cortex and the cathode over the left dorsolateral prefrontal cortex, positioned at F4 and F3, respectively, according to the International 10/20 Electrode Placement System. The current intensity will be set to 2 milliamperes (mA) for 20 minutes over five consecutive days.
  Other Names: transcranial Direct Current Stimulation
  Arms: tDCS Sham group; tDCS True Modulation
Device: tVNS — For true tVNS stimulation, the technique will be performed with the electrodes positioned on the upper concha of the left ear, using gel for better current distribution.
  Other Names: transcutaneous Vagus Nerve Stimulation
  Arms: tVNS Sham; tVNS True

SUMMARY:
This clinical trial aims to determine if Transcranial electrical stimulation by direct current (tDCS) and transauricular Vagus Nerve Stimulation (tVNS) treatments are effective in reducing stress symptoms, distress and improving sleep quality in adults. The main questions it aims to answer are:

* Determine if tDCS effectively reduces the intensity of stress symptoms in adults.
* Determine if tDCS is effective in reducing levels of distress in adults.
* Determine if tDCS is effective in improving sleep quality.
* Determine if tVNS is effective in reducing the intensity of stress symptoms in adults.
* Determine if tVNS is effective in reducing levels of distress in adults.
* Determine if tVNS is effective in improving sleep quality.

DETAILED DESCRIPTION:
Stress is a disorder that significantly impacts the lives of affected individuals. Pharmacological treatment has limitations, justifying the search for non-pharmacological interventions. tDCS is a technique that modulates neuronal excitability and has shown promising results in various disorders.

Psychological stress affects a wide range of brain functions and poses risks for many mental disorders. However, effective therapies to alleviate or reverse its deleterious effects are lacking. Given that the pathophysiology of stress involves brain regions such as the prefrontal cortex, central amygdaloid nucleus, amygdala, medial amygdaloid nucleus, and ventral hippocampus, thus making the condition complex, there is a need for studies evaluating the effects of this intervention. We aim to contribute to the understanding of the role of tDCS and tVNS in managing stress.

Before participating in this research, volunteers will receive all information related to the study's objectives and methodological procedures. After agreeing to participate, they will sign the Informed Consent Form.

Study Location Patients will be selected following an evaluation based on inclusion and exclusion criteria and referred to the Clinic School of the Federal University of Alfenas (MG/Brazil), at the Laboratory of Neuroscience, Neuromodulation, and Pain Study (LANNED), located in the city of Alfenas, Minas Gerais, and at the Neuromodulation and Pain Unit (UNP) by the Egas Moniz Center for Interdisciplinary Research (CiiEM) of the Egas Moniz School of Health and Science, in the municipality of Almada, Setúbal - Portugal.

The design of the double-blind randomized clinical trial will be conducted, ensuring that participants are randomly assigned to experimental and sham groups and that the researcher applying the technique and the participants will not be aware of the allocation. The protocol will consist of 5 consecutive sessions of 20 minutes each. Data related to the anamnesis, ISSL, PSS-10, and PSQI will be evaluated at five different time points (Figure 1): before the intervention (T0), immediately after the end of the intervention (T1), and four weeks (T2) after the intervention ends (follow-up), following the CONSORT/2010 recommendations.

ELIGIBILITY:
Inclusion Criteria:

* individuals previously diagnosed with stress.
* Obtain a score above 4 on the Lipp Adult Stress Symptom Inventory (ISSL);
* Must be able to read and understand the purpose of the research and respond to the assessment instruments.
* Must acknowledge and agree with the informed consent form.

Exclusion Criteria:

* smokers;
* be pregnant;
* initiation and/or change in psychotropic drug dosage in the last three months;
* use of anxiolytics or antidepressants;
* substance dependence;
* history of dizziness or seizures;
* signs of severity and/or indications for hospitalization or psychotherapy;
* diagnosis of depression; diagnosis of anxiety; bipolar mood disorder with depressive, manic, or hypomanic symptoms in the past year;
* schizophrenia or other psychotic disorders;
* autism;
* diagnosis of epilepsy or use of anticonvulsants;
* contraindications for tDCS (metal implants, tumor, previous brain surgery, significant cranioencephalic anatomical alterations);
* contraindications for non-invasive vagus nerve stimulation (cochlear implant, ear plastic surgery, ear malformation);
* adverse effects detected in the group treated with tDCS and tVNS, including itching, tingling, headache, burning sensation, and discomfort.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Stress Symptoms assessment | From enrollment to follow up at 1 month
  Stress will be assessed using self reported Lipp's Inventory of Stress Symptoms for Adults (LISS). The LISS consists of a questionnaire that assesses physical and psychological symptoms of stress across three time frames: alert (ranging from 0 to 15), resistance (ranging from 0 to 15), quasi-exhaustion or exhaustion (ranging from 0 to 23). Higher scores mean a worse outcome.
Perceived Stress assessment | From enrollment to follow up at 1 month
  Perceived Stress will be assessed using the Perceived Stress Scale (PSS-10). The test ranges from 0 (min) to 40 (max). Higher scores mean a a worst outcome.

SECONDARY OUTCOMES:
Distress Assessment | From enrollment to followup at 1 month
  Distress will be assessed using the Kessler Psychological Distress Scale (K10). the scale range is from 10 (min) to 50 (max). Higher scores mean a worse outcome.
Sleep Quality | From enrollment to follow up at 1 month
  Stress will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The global PSQI score ranges from 0 to 21. Higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Egas Moniz Scholl Of Health and Science, Almada, Setúbal District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunoni AR, Nitsche MA, Bolognini N, Bikson M, Wagner T, Merabet L, Edwards DJ, Valero-Cabre A, Rotenberg A, Pascual-Leone A, Ferrucci R, Priori A, Boggio PS, Fregni F. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. Brain Stimul. 2012 Jul;5(3):175-195. doi: 10.1016/j.brs.2011.03.002. Epub 2011 Apr 1. PMID 22037126
- [Background] Alyan E, Saad NM, Kamel N, Yusoff MZ, Zakariya MA, Rahman MA, Guillet C, Merienne F. Frontal Electroencephalogram Alpha Asymmetry during Mental Stress Related to Workplace Noise. Sensors (Basel). 2021 Mar 11;21(6):1968. doi: 10.3390/s21061968. PMID 33799722
- [Background] Loftus AM, Yalcin O, Baughman FD, Vanman EJ, Hagger MS. The impact of transcranial direct current stimulation on inhibitory control in young adults. Brain Behav. 2015 May;5(5):e00332. doi: 10.1002/brb3.332. Epub 2015 Mar 19. PMID 25874165